## ADHESIVE DEVICES VERSUS ELASTIC DEVICES FOR URINARY CATHETER SECUREMENT IN CRITICALLY ILL PATIENTS. EXPERIMENTAL STUDY

STATISTICAL ANALYSES PLAN

Code: IIBSP-DAE-2025-22 Version: 1. Date: 18/02/2025

## **Data Analysis**

A descriptive analysis of the variables will be performed. Qualitative variables will be described using frequencies and percentages, and quantitative variables using mean and standard deviation or median and 25th and 75th percentiles, depending on their distribution. The Kolmogorov-Smirnov test will be used to assess the normality of continuous variables. Subsequently, a bivariate analysis will be conducted according to the study objectives.

To compare a variable between two independent groups, the Student's t-test will be used for normally distributed variables, the Mann-Whitney U test for non-normal variables, and the Chi-square test or Fisher's exact test for two qualitative variables.

Additionally, variables that show a statistically significant or clinically relevant association will be included in a multiple logistic regression model to identify factors independently associated with urinary meatus lesions and catheter-associated urinary tract infections (CAUTI). A significance level of p < 0.05 will be established.

Code: IIBSP-DAE-2025-22 Version: 1. Date: 18/02/2025